CLINICAL TRIAL: NCT00511888
Title: Effects of Nebivolol Versus Carvedilol in Hypertensive Patients With Chronic Heart Failure
Brief Title: Nebivolol Versus Carvedilol in Patients With Heart Failure
Status: Terminated | Type: Observational
Why Stopped: is finish
Sponsor: IRCCS San Raffaele (Other)
Other Study IDs: 001-07
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-08

CONDITIONS: Chronic Heart Failure; Hypertension
Keywords: chronic heart failure; hypertension; beta blockers
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
BACKGROUND Beta-blockers improve left ventricular (LV) systolic function and prognosis in patients with chronic heart failure. Both carvedilol and nebivolol have hemodynamic and clinical benefits in chronic heart failure (CHF), but it is unknown whether their pleiotropic properties may play a role in different subgroups of patients with CHF.

OBJECTIVE: To compare the effects of nebivolol and carvedilol on LV function and clinical outcome in patients with chronic heart failure and reduced LV systolic function.

METHODS: 160 hypertensive CHF patients, LV ejection fraction (EF) 40% and in New York Heart Association (NYHA) functional class II or III were randomly assigned to receive carvedilol or nebivolol therapy for 24 months. At baseline and after 24 months of treatment, all patients underwent clinical evaluation: echocardiogram and 6-minute walking test.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction (LVEF) < 40%;
* symptomatic heart failure with functional New York Heart Association (NYHA) class II or III;
* arterial hypertension with systolic blood pressure >140 mmHg and diastolic blood pressure >85 mmHg;
* clinical stability without hospital admission for heart failure in the previous 3 months.

Exclusion Criteria:

* history of asthma or severe chronic obstructive pulmonary disease;
* severe liver or kidney diseases;
* second-degree or third degree heart block without a permanent pacemaker,
* sick sinus syndrome, heart rate <60 beat/min, systolic blood pressure <90 mmHg.

Ages: 53 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: giuseppe rosano, md, Study Director — IRCCS san Raffaele Cardiovascular Research Unit
Locations (1):
- IRCCS San Raffaele, Rome, rome, Italy